CLINICAL TRIAL: NCT03910907
Title: Comparison of Current Standard of Care Versus the Australian Guidelines for Management of Mycoplasma Genitalium Infections Among Men Being Treated for Non-gonococcal Urethritis
Brief Title: Comparison of Standard of Care Guidelines for Mycoplasma Genitalium Infections Among Men With Non-gonococcal Urethritis
Status: Terminated | Type: Observational
Why Stopped: Covid
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Barbara Van Der Pol, Primary Investigator, University of Alabama at Birmingham
Other Study IDs: IRB-300003178
Record Dates: First submitted 2019-04-08; First posted 2019-04-10 (Actual); Last update posted 2023-06-02 (Actual); Status verified 2023-06

CONDITIONS: Mycoplasma Genitalium Infection
Keywords: mycoplasma genitalium; urethritis; NGU; treatment
MeSH Terms: conditions — Urethritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Residual urine samples will be retained
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (2):
- Standard of care: Men treated for mycoplasma according to standard of care
  Interventions: Drug: Comparison of two standard of care regimens
- Standard of care plus: Men treated for mycoplasma according to standard of care with regimen selected based on laboratory detection of resistance markers
  Interventions: Drug: Comparison of two standard of care regimens

INTERVENTIONS:
Drug: Comparison of two standard of care regimens — Treatment according to results of laboratory detection of resistance markers

SUMMARY:
The purpose of this protocol is to determine the difference in clearance of Mycoplasma genitalium (MG) when using the Australian management protocol versus the current Centers of Disease Control (CDC) treatment guidelines for US standard of care (SOC), to determine the proportion of men from the Deep South, with NGU attributable to MG, and to determine the proportion of MG cases that harbor the macrolide-resistance associated with mutation.

DETAILED DESCRIPTION:
Mycoplasma genitalium (MG) has been associated with non-gonococcal urethritis (NGU) in many populations and the prevalence of MG strains with macrolide-resistance associated gene mutations is increasing . While no MG diagnostic assays have FDA clearance in the United States (US), treatment for NGU is primarily focused on managing potential infection with Chlamydia trachomatis (CT) using single dose 1 gm Azithromycin (a macrolide class of drug). Without testing for MG that might alter NGU treatment strategies, the current paradigm may be contributing to selective pressure resulting in increased macrolide resistance in MG. In Australia, awareness of the prevalence of MG and macrolide resistance-associated mutations has been facilitated by an approved diagnostic test manufactured by SpeeDx. Ltd. As a result of the epidemiologic information generated by this diagnostic tool [MG ResistancePlus (MRP) Assay], the Australian Sexual Health Alliance, who publish the Australian Sexually Transmitted Infection (STI) Management Guidelines for Use in Primary Care, have revised the management of men with NGU and MG infection. The new management guidelines include initial treatment of NGU with doxycycline, and concomitant testing for MG and macrolide resistance, with subsequent treatment for MG infected patients according to resistance results. We propose using the MRP assay in a population of men with NGU to determine the clinical impact of the Australian treatment strategy compared to the current standard of care for NGU on clearance of MG infection.

ELIGIBILITY:
Inclusion Criteria:

* Presenting with symptoms of urethritis (dysuria and/or urethral discharge)

Exclusion Criteria:

* Non-English speaking

Ages: 18 Years to 99 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Men with non-gonoccocal
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2019-11-19 (Actual); Primary Completion 2020-03-20 (Actual); Study Completion 2020-03-20 (Actual)

PRIMARY OUTCOMES:
Participants with Molecular Clearance | 90 days
  DNA negative for mycoplasma

SECONDARY OUTCOMES:
Positive Participants with Macrolide-Resistant Mycoplasma | 90 days
  DNA positive for macrolide-resistant mycoplasma

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Van Der Pol, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- UAB, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No